CLINICAL TRIAL: NCT01396707
Title: A Phase II Study of Trastuzumab in Combination With Capecitabine and Oxaliplatin (XELOX) in Patients With Advanced Gastric Cancer
Brief Title: Trastuzumab in Combination With Capecitabine and Oxaliplatin(XELOX) in Patients With Advanced Gastric Cancer(AGC): Her+XELOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC1101
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Metastatic or Recurrent Gastric Adenocarcinoma; Her-2 Positive Gastric Cancer
Keywords: HER2; Trastuzumab; XELOX; PHASE 2
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Trastuzumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Herceptin+XELOX (Experimental)
  Interventions: Drug: Herceptin+XELOX

INTERVENTIONS:
Drug: Herceptin+XELOX — Each 3-weekly cycle, with chemotherapy given for 6 cycles, and trastuzumab continued even after completion of the combination chemotherapy until disease progression
  * Trastuzumab: 8 mg/kg i.v. loading dose on day 1, followed by 6 mg/kg i.v.infusion every 3 weeks
  * Capecitabine: 1000 mg/m2 oral twice daily for 14 days every 3 weeks (from evening on day 1 to morning on day 15)
  * Oxaliplatin 130 mg/m2 i.v. on day 1
  Other Names: Trastuzumab; Capecitabine; Oxaliplatin

SUMMARY:
This is an open-label, multicentre, prospective phase II trial designed to evaluate the efficacy and safety of trastuzumab in combination with capecitabine and oxaliplatin as first-line therapy in patients with recurrent and/or metastatic HER2 positive adenocarcinoma of the stomach or gastro-oesophageal junction.

DETAILED DESCRIPTION:
Patients will be administered 6 cycles of combination chemotherapy, unless withdrawn earlier due to unacceptable toxicity, disease progression, or consent withdrawal. Patients will continue to be treated with trastuzumab alone until disease progression, unacceptable toxicity or consent withdrawal after finishing a maximum 6 cycles of combination chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the stomach or gastro-oesophageal junction with inoperable locally advanced or recurrent and/or metastatic disease, not amenable to curative therapy.
2. Measurable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST), assessed using imaging techniques (CT or MRI).
3. HER2 positive tumour (primary tumour or metastasis) defined as either IHC2+ and FISH+ or IHC3+ according to the gastric cancer scoring system for HER2
4. ECOG Performance status 0, 1 or 2
5. Life expectancy of at least 3 months.
6. Male or female. Age over 20 year.
7. Signed informed consent.

Exclusion Criteria:

1. Previous chemotherapy for advanced/metastatic disease (prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the study; adjuvant/neoadjuvant therapy with platinum is not allowed).
2. Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome (e.g. patients with partial or total gastrectomy can enter the study, but not those with a jejunostomy tube).
3. Patients with active (significant or uncontrolled) gastrointestinal bleeding.
4. Residual relevant toxicity resulting from previous therapy (with the exception of alopecia), e.g. neurological toxicity over grade 2 NCI-CTCAE.
5. Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma.
6. Neutrophil count < 1.5 × 109/L, or platelet count < 100 × 109/L.
7. Serum bilirubin > 1.5 × upper limit of normal (ULN); or, AST or ALT > 2.5 × ULN (or > 5 × ULN in patients with liver metastases); or, alkaline phosphatase > 2.5 × ULN (or > 5 × ULN in patients with liver metastases, or > 10 × ULN in patients with bone but no liver metastases); or, albumin < 25 g/L.
8. Creatinine clearance < 60 mL/min. Other Study Drug-Related Exclusion Criteria
9. History of documented congestive heart failure; angina pectoris requiring medication; evidence of transmural myocardial infarction on ECG; poorly controlled hypertension (systolic BP > 180 mmHg or diastolic BP > 100 mmHg); clinically significant valvular heart disease; or high risk uncontrollable arrhythmias.
10. Baseline LVEF < 50% (measured by echocardiography or MUGA).
11. Patients with dyspnea at rest due to complications of advanced malignancy or other disease, or who require supportive oxygen therapy.
12. Patients receiving chronic or high dose corticosteroid therapy. (Inhaled steroids and short courses of oral steroids for anti-emesis or as an appetite stimulant are allowed).
13. Clinically significant hearing abnormality.
14. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
15. History or clinical evidence of brain metastases.
16. Serious uncontrolled systemic intercurrent illness, e.g. infections or poorly controlled diabetes.
17. Positive serum pregnancy test in women of childbearing potential.
18. Subjects with reproductive potential not willing to use an effective method of contraception.
19. Received any investigational drug treatment within 4 weeks of start of study treatment.
20. Radiotherapy within 4 weeks of start of study treatment (2 week interval allowed if palliative radiotherapy given to bone metastatic site peripherally and patient recovered from any acute toxicity).
21. Major surgery within 4 weeks of start of study treatment, without complete recovery.
22. History of HIV infection, Patients with known active infection with HBV, or HCV.
23. Known hypersensitivity to any of the study drugs.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 1 year
  To evaluate the overall response rate for patients treated with trastuzumab combinated with capecitabine plus oxaliplatin.

SECONDARY OUTCOMES:
Duration of response | 1 year
Time to progression | 1 year
Progression free survival | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parkin DM, Pisani P, Ferlay J. Global cancer statistics. CA Cancer J Clin. 1999 Jan-Feb;49(1):33-64, 1. doi: 10.3322/canjclin.49.1.33. PMID 10200776
- [Background] Murad AM, Santiago FF, Petroianu A, Rocha PR, Rodrigues MA, Rausch M. Modified therapy with 5-fluorouracil, doxorubicin, and methotrexate in advanced gastric cancer. Cancer. 1993 Jul 1;72(1):37-41. doi: 10.1002/1097-0142(19930701)72:13.0.co;2-p. PMID 8508427
- [Background] Glimelius B, Ekstrom K, Hoffman K, Graf W, Sjoden PO, Haglund U, Svensson C, Enander LK, Linne T, Sellstrom H, Heuman R. Randomized comparison between chemotherapy plus best supportive care with best supportive care in advanced gastric cancer. Ann Oncol. 1997 Feb;8(2):163-8. doi: 10.1023/a:1008243606668. PMID 9093725
- [Background] Pyrhonen S, Kuitunen T, Nyandoto P, Kouri M. Randomised comparison of fluorouracil, epidoxorubicin and methotrexate (FEMTX) plus supportive care with supportive care alone in patients with non-resectable gastric cancer. Br J Cancer. 1995 Mar;71(3):587-91. doi: 10.1038/bjc.1995.114. PMID 7533517
- [Background] Kim NK, Park YS, Heo DS, Suh C, Kim SY, Park KC, Kang YK, Shin DB, Kim HT, Kim HJ, et al. A phase III randomized study of 5-fluorouracil and cisplatin versus 5-fluorouracil, doxorubicin, and mitomycin C versus 5-fluorouracil alone in the treatment of advanced gastric cancer. Cancer. 1993 Jun 15;71(12):3813-8. doi: 10.1002/1097-0142(19930615)71:123.0.co;2-5. PMID 8508349
- [Background] Ohtsu A, Shimada Y, Shirao K, Boku N, Hyodo I, Saito H, Yamamichi N, Miyata Y, Ikeda N, Yamamoto S, Fukuda H, Yoshida S; Japan Clinical Oncology Group Study (JCOG9205). Randomized phase III trial of fluorouracil alone versus fluorouracil plus cisplatin versus uracil and tegafur plus mitomycin in patients with unresectable, advanced gastric cancer: The Japan Clinical Oncology Group Study (JCOG9205). J Clin Oncol. 2003 Jan 1;21(1):54-9. doi: 10.1200/JCO.2003.04.130. PMID 12506170
- [Background] Mackean M, Planting A, Twelves C, Schellens J, Allman D, Osterwalder B, Reigner B, Griffin T, Kaye S, Verweij J. Phase I and pharmacologic study of intermittent twice-daily oral therapy with capecitabine in patients with advanced and/or metastatic cancer. J Clin Oncol. 1998 Sep;16(9):2977-85. doi: 10.1200/JCO.1998.16.9.2977. PMID 9738566
- [Background] Kim TW, Kang YK, Ahn JH, Chang HM, Yook JH, Oh ST, Kim BS, Lee JS. Phase II study of capecitabine plus cisplatin as first-line chemotherapy in advanced gastric cancer. Ann Oncol. 2002 Dec;13(12):1893-8. doi: 10.1093/annonc/mdf323. PMID 12453857
- [Background] Kang YK, Kang WK, Shin DB, Chen J, Xiong J, Wang J, Lichinitser M, Guan Z, Khasanov R, Zheng L, Philco-Salas M, Suarez T, Santamaria J, Forster G, McCloud PI. Capecitabine/cisplatin versus 5-fluorouracil/cisplatin as first-line therapy in patients with advanced gastric cancer: a randomised phase III noninferiority trial. Ann Oncol. 2009 Apr;20(4):666-73. doi: 10.1093/annonc/mdn717. Epub 2009 Jan 19. PMID 19153121
- [Background] Mamenta EL, Poma EE, Kaufmann WK, Delmastro DA, Grady HL, Chaney SG. Enhanced replicative bypass of platinum-DNA adducts in cisplatin-resistant human ovarian carcinoma cell lines. Cancer Res. 1994 Jul 1;54(13):3500-5. PMID 8012973
- [Background] Schmidt W, Chaney SG. Role of carrier ligand in platinum resistance of human carcinoma cell lines. Cancer Res. 1993 Feb 15;53(4):799-805. PMID 8428361
- [Background] Andre T, Bensmaine MA, Louvet C, Francois E, Lucas V, Desseigne F, Beerblock K, Bouche O, Carola E, Merrouche Y, Morvan F, Dupont-Andre G, de Gramont A. Multicenter phase II study of bimonthly high-dose leucovorin, fluorouracil infusion, and oxaliplatin for metastatic colorectal cancer resistant to the same leucovorin and fluorouracil regimen. J Clin Oncol. 1999 Nov;17(11):3560-8. doi: 10.1200/JCO.1999.17.11.3560. PMID 10550155
- [Background] Royce ME, Hoff PM, Pazdur R. Progress in colorectal cancer chemotherapy: how far have we come, how far to go? Drugs Aging. 2000 Sep;17(3):201-16. doi: 10.2165/00002512-200017030-00004. PMID 11043819
- [Background] Eriguchi M, Nonaka Y, Yanagie H, Yoshizaki I, Takeda Y, Sekiguchi M. A molecular biological study of anti-tumor mechanisms of an anti-cancer agent Oxaliplatin against established human gastric cancer cell lines. Biomed Pharmacother. 2003 Nov;57(9):412-5. doi: 10.1016/s0753-3322(03)00027-1. PMID 14652166
- [Background] Cassidy J, Misset JL. Oxaliplatin-related side effects: characteristics and management. Semin Oncol. 2002 Oct;29(5 Suppl 15):11-20. doi: 10.1053/sonc.2002.35524. PMID 12422304
- [Background] Park YH, Lee JL, Ryoo BY, Ryu MH, Yang SH, Kim BS, Shin DB, Chang HM, Kim TW, Yuh YJ, Kang YK. Capecitabine in combination with Oxaliplatin (XELOX) as a first-line therapy for advanced gastric cancer. Cancer Chemother Pharmacol. 2008 Apr;61(4):623-9. doi: 10.1007/s00280-007-0515-7. Epub 2007 May 24. PMID 17522863
- [Background] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Background] Al-Batran SE, Hartmann JT, Probst S, Schmalenberg H, Hollerbach S, Hofheinz R, Rethwisch V, Seipelt G, Homann N, Wilhelm G, Schuch G, Stoehlmacher J, Derigs HG, Hegewisch-Becker S, Grossmann J, Pauligk C, Atmaca A, Bokemeyer C, Knuth A, Jager E; Arbeitsgemeinschaft Internistische Onkologie. Phase III trial in metastatic gastroesophageal adenocarcinoma with fluorouracil, leucovorin plus either oxaliplatin or cisplatin: a study of the Arbeitsgemeinschaft Internistische Onkologie. J Clin Oncol. 2008 Mar 20;26(9):1435-42. doi: 10.1200/JCO.2007.13.9378. PMID 18349393
- [Background] Hofmann M, Stoss O, Shi D, Buttner R, van de Vijver M, Kim W, Ochiai A, Ruschoff J, Henkel T. Assessment of a HER2 scoring system for gastric cancer: results from a validation study. Histopathology. 2008 Jun;52(7):797-805. doi: 10.1111/j.1365-2559.2008.03028.x. Epub 2008 Apr 18. PMID 18422971